CLINICAL TRIAL: NCT06832826
Title: Challenges in Colonic Polypectomy and Endoscopic Mucosal Resection in Cirrhotic Patients With Portal Hypertension: Single-Center Experience
Brief Title: Colonic Polypectomy in Cirrhotic Patients With Portal Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Other Study IDs: ZU-IRB#851/1-Dec-2024
Record Dates: First submitted 2025-01-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Liver Cirrhosis; Portal Hypertension Related to Cirrhosis; Polyp of Colon; Polypectomy
Keywords: colonic polyp; polypectomy; portal hypertension; post-polypectomy bleeding
MeSH Terms: conditions — Liver Cirrhosis; Colonic Polyps; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver cirrhosis patients with portal hypertension and colonic polyps: Colonic polypectomy

SUMMARY:
The goal of this retrospective cohort study is to evaluate the risk of post-polypectomy bleeding following the colonoscopy resection of lower gastrointestinal polyps in patients with liver cirrhosis with portal hypertension. The main question it aims to answer is:

Does the risk of bleeding increase after colonoscopy polypectomy in patients with liver cirrhosis with portal hypertension?

Participants will be subjected to polypectomy of any colonic polyps.

ELIGIBILITY:
Inclusion Criteria:

* All liver cirrhosis patients with portal hypertension and colonic polyps

Exclusion Criteria:

* Patients with platelet count less than 50,000/µL.
* Patients with hemoglobin levels less than 8 g/dL.
* Prothrombin Time more than 20 seconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver cirrhosis patients with evidence of portal hypertension
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Immediate post polypectomy bleeding (IPPB) | During procedure
Delayed post polypectomy bleeding (DPPB) | 24 hours to 14 days

SECONDARY OUTCOMES:
Type of polyps in patients with liver cirrhosis and portal hypertension | 14 days
  Using the Paris classification system for polyps

OTHER OUTCOMES:
Prediction of risk of post polypectomy bleeding | 6 months
  Using the updated Endoscopic Resection Group of the Spanish Society of Endoscopy model and the Australian Colonic Endoscopic Resection model

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Study Director — Zagazig University
Locations (1):
- Zagazig University Hospital, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee S, Park SJ, Cheon JH, Kim TI, Kim WH, Kang DR, Hong SP. Child-Pugh score is an independent risk factor for immediate bleeding after colonoscopic polypectomy in liver cirrhosis. Yonsei Med J. 2014 Sep;55(5):1281-8. doi: 10.3349/ymj.2014.55.5.1281. PMID 25048486
- [Result] Amarapurkar AD, Amarapurkar D, Choksi M, Bhatt N, Amarapurkar P. Portal hypertensive polyps: distinct entity. Indian J Gastroenterol. 2013 May;32(3):195-9. doi: 10.1007/s12664-013-0324-3. Epub 2013 Mar 20. PMID 23512212
- [Result] Jeon JW, Shin HP, Lee JI, Joo KR, Pack KM, Cha JM, Park JJ, Lim JU, Lim K. The risk of postpolypectomy bleeding during colonoscopy in patients with early liver cirrhosis. Surg Endosc. 2012 Nov;26(11):3258-63. doi: 10.1007/s00464-012-2334-0. Epub 2012 May 31. PMID 22648106
- [Result] Hui AJ, Wong RM, Ching JY, Hung LC, Chung SC, Sung JJ. Risk of colonoscopic polypectomy bleeding with anticoagulants and antiplatelet agents: analysis of 1657 cases. Gastrointest Endosc. 2004 Jan;59(1):44-8. doi: 10.1016/s0016-5107(03)02307-1. PMID 14722546
- [Result] Gibbs DH, Opelka FG, Beck DE, Hicks TC, Timmcke AE, Gathright JB Jr. Postpolypectomy colonic hemorrhage. Dis Colon Rectum. 1996 Jul;39(7):806-10. doi: 10.1007/BF02054448. PMID 8674375
- [Result] Rosen L, Bub DS, Reed JF 3rd, Nastasee SA. Hemorrhage following colonoscopic polypectomy. Dis Colon Rectum. 1993 Dec;36(12):1126-31. doi: 10.1007/BF02052261. PMID 8253009
- [Result] Giannini EG, Greco A, Marenco S, Andorno E, Valente U, Savarino V. Incidence of bleeding following invasive procedures in patients with thrombocytopenia and advanced liver disease. Clin Gastroenterol Hepatol. 2010 Oct;8(10):899-902; quiz e109. doi: 10.1016/j.cgh.2010.06.018. Epub 2010 Jun 30. PMID 20601131
- [Result] Cocero N, Bezzi M, Martini S, Carossa S. Oral Surgical Treatment of Patients With Chronic Liver Disease: Assessments of Bleeding and Its Relationship With Thrombocytopenia and Blood Coagulation Parameters. J Oral Maxillofac Surg. 2017 Jan;75(1):28-34. doi: 10.1016/j.joms.2016.08.033. Epub 2016 Sep 2. PMID 27677683
- [Result] Tripodi A. Hemostasis abnormalities in cirrhosis. Curr Opin Hematol. 2015 Sep;22(5):406-12. doi: 10.1097/MOH.0000000000000164. PMID 26203733
- [Result] Mucino-Bermejo J, Carrillo-Esper R, Mendez-Sanchez N, Uribe M. Thrombosis and hemorrhage in the critically ill cirrhotic patients: five years retrospective prevalence study. Ann Hepatol. 2015 Jan-Feb;14(1):93-8. PMID 25536646